CLINICAL TRIAL: NCT04307147
Title: Study Evaluating Vinorelbine Plus Capecitabine in the Treatment of Luminal B Breast Cancer Patients After Neoadjuvant Chemotherapy
Brief Title: NX in Luminal B Breast Cancer Patients After Neoadjuvant Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fudan University
Record Dates: First submitted 2020-03-08; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NX (vinorelbine and capecitabine ) (Experimental): Standard therapy plus NX chemotherapy for 4 cycles, (vinorelbine 25 mg/m² d1,8 and capecitabine 1250 mg/m² d1-14, every 3 weeks)
  Interventions: Drug: Capecitabine; Drug: Vinorelbine
- Control group (No Intervention): Standard therapy

INTERVENTIONS:
Drug: Capecitabine — Oral capecitabine (at a dose of 1250 mg/m², twice per day, on days 1 to 14) every 3 weeks for 4 cycles.
  Arms: NX (vinorelbine and capecitabine )
Drug: Vinorelbine — Intravenous vinorelbine (at a dose of 25 mg/m² on day 1, day 8) every 3 weeks for 4 cycles.
  Arms: NX (vinorelbine and capecitabine )

SUMMARY:
This is a prospective, randomized, open-lable phase III clinical trial evaluating the effectiveness and safety of vinorelbine plus capecitabine as adjuvant treatment for non-pCR Luminal B breast cancer patients after standard neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
This is a prospective ,randomized, open-lable phase III clinical trial evaluating the effectiveness and safety of vinorelbine plus capecitabine as adjuvant treatment for non-pCR Luminal B breast cancer patients after standard neoadjuvant chemotherapy. Non-pCR Luminal B patients who completed 6-8 cycles of standard neoadjuvant chemotherapy will be included in this study and receive 4 cycles of NX regimen chemotherapy for 4 cycles (vinorelbine 25 mg/m² d1,8 and capecitabine 1250 mg/m² d1-14, every 3 weeks) or not. the investigator's primary endpoint is disease free survival (DFS). Secondary end points include overall survival (OS), recurrence free survival (RFS), distant disease free survival (DDFS)rates and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years old
* Patients with histologically confirmed unilateral invasive ductal
* carcinoma(according to WHO histologically type)
* Tumor clinical staged as IIB-IIIB before neoadjuvant chemotherapy (according to the 7th AJCC edition).
* After standard treatment (6-8 cycles) of neoadjuvant chemotherapy (plan formulated by the attending doctor, including anthracycline and paclitaxel drugs, must not contain platinum), assessed by the surgery, the original site for non - pCR (MP class 1-4) or lymph nodes are still positive for patients.
* Luminal B breast cancer defined as positive oestrogen and/or progesterone receptors, a negative HER2 defined as negative ISH test or an IHC status of 0 or 1+ as per local laboratory testing and a Ki67 > 14%.
* No evidence of distant metastasis in the clinical or radiological aspects of preoperative. examination,that is M0.
* Patients without peripheral neuropathy or I peripheral neurotoxicity.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤1.
* Patients recovered well after surgery, at least 1 weeks after the operation.
* Adequate marrow: White blood cells count≥3000/μL,neutrophil count ≥1500/μL, hemoglobin ≥9g/dL and platelet count ≥75000/μL.
* Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) ≤ 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤ 2.5×ULN, and bilirubin ≤ 1.5ULN.
* Adequate renal function: Serum creatinine ≤ 1.5ULN.
* Contraception during the treatment of child-bearing women.
* Adequate cardiac function :Left ventricular ejection fraction (LVEF) > 50%.
* Patients must be informed of the investigational nature of this study and give written informed consent.
* Patients without serious heart, lung, liver, kidney and other important organs disease history.
* Patients have good compliance.

Exclusion Criteria:

* Patients with bilateral breast cancer or carcinoma in situ(DCIS/LCIS).
* Metastasis of any part except axillary lymph nodes.
* Clinical or imaging suspicion of the contralateral breast is malignant but not confirmed, requiring biopsy.
* There have been malignant tumors (except for basal cell carcinoma and carcinoma in situ of cervix) in the last five years, including breast cancer.
* Patients have been enrolled in other clinical trials.
* Patients with severe systemic illnesses and/or uncontrolled infections are unable to join the study.
* Patients with severe cardio-cerebrovascular disorders (e.g., unstable angina pectoris, chronic heart failure, uncontrollable hypertension >160/100mmgh, myocardial infarction or cerebrovascular accident) in the first 6 months of randomization.
* Pregnant lactating women (child-bearing women must be negative for pregnancy test within 14 days prior to first delivery, if positive, the pregnancy should be excluded by ultrasound.)
* Child-bearing women who are unwilling to take effective contraceptive measures in the course of research.
* Patients with mental illness, cognitive impairment, inability to understand test protocols and side effects, and those who fail to complete the trial programme and follow-up work (a systematic assessment is required before the trial).
* Persons without personal freedom and independent civil capacity.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2018-07-03 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 5-year
  The length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer

SECONDARY OUTCOMES:
Overall survival | 5-year
  Overall survival is calculated from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital/ Institute, Fudan University, Shanghai, Shanghai Municipality, China